CLINICAL TRIAL: NCT05453851
Title: Total Pancreatectomy With Islet Cell Autotransplantation in Patients With Benign Pancreatic Neoplasms: A Pilot Study
Brief Title: A Surgical Procedure (Total Pancreatectomy) With a Transplant Procedure (Islet Cell Autotransplantation) for the Treatment of Chronic Pancreatitis and Benign Pancreatic Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brett C. Sheppard, M.D., FACS, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00023937; NCI-2022-05134 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023937 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Benign Pancreatic Neoplasm; Chronic Pancreatitis; Recurrent Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Pancreatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pancreatectomy, autologous islet cell transplant) (Experimental): Patients undergo total pancreatectomy and autologous islet cell transplant IV over 15-60 minutes on day 1.
  Interventions: Procedure: Pancreatectomy; Other: Quality-of-Life Assessment; Other: Treatment Planning

INTERVENTIONS:
Procedure: Pancreatectomy — Undergo pancreatectomy
  Other Names: Excision of the Pancreas; Pancreas Excision
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Treatment Planning — Undergo IV autologous islet cell transplant

SUMMARY:
This phase I/II trial assesses the safety and effectiveness of total pancreatectomy with islet cell autotransplantation for the treatment of patients with long-term pancreatic inflammation (chronic pancreatitis) and non-cancerous (benign) pancreatic tumors. Total removal of the pancreas (pancreatectomy) can be used to treat chronic pancreatitis, but it may result in diabetes. An islet cell autotransplantation involves removing cells from a patient's pancreas (the islet cells) and infusing them into the liver. Islet cells are responsible for producing hormones like insulin, reducing the occurrence of diabetes in patients undergoing total pancreatectomy. Total pancreatectomy with autologous islet cell transplant is an accepted and Food and Drug Administration-approved treatment for patients with chronic pancreatitis. However, patients with chronic pancreatitis and pancreatic tumors have historically not been candidates for this procedure due to concerns of spreading potentially cancerous cells to other parts of the body. This clinical trial evaluates the safety and effectiveness of this treatment in patients with chronic pancreatitis and benign pancreatic tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the oncologic safety of total pancreatectomy with islet cell autotransplantation (TPIAT) in chronic pancreatitis patients with benign pancreatic neoplasms.

SECONDARY OBJECTIVES:

I. To evaluate postoperative insulin requirements in patients with presumed benign pancreatic neoplasms undergoing TPIAT.

II. To evaluate postoperative opiate requirements in patients with presumed benign pancreatic neoplasms undergoing TPIAT.

III. To evaluate the postoperative survival of patients with presumed benign pancreatic neoplasms undergoing TPIAT.

EXPLORATORY OBJECTIVES:

I. To evaluate quality of life outcomes in patients undergoing TPIAT with presumed benign pancreatic neoplasms.

II. To evaluate subjective pain-related outcomes in patients undergoing TPIAT with presumed benign pancreatic neoplasms.

OUTLINE:

Patients undergo total pancreatectomy and autologous islet cell transplant intravenously (IV) over 15-60 minutes on day 1.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative (LAR) must provide written informed consent before any study-specific procedures or interventions are performed
* Age>= 18 years. Both men and women and members of all races and ethnic groups will be included. Gender-nonconforming and gender-fluid individuals as members of the general population will also be included
* Participants must have adequate islet cell function (non-diabetic or C-peptide positive)
* Participants must be indicated for total surgical resection of the pancreas for chronic pancreatitis-associated pain meeting eligibility criteria for TPIAT per University of Minnesota Criteria as defined by all of the following

  * Chronic abdominal pain of > 6-month duration with at least one of the following:

    * Pancreatic calcification on computed tomography (CT) scan
    * At least two of the following:

      * Definite of suggestive diagnosis of chronic pancreatitis on endoscopic ultrasound
      * Ductal or parenchymal abnormalities compatible with chronic pancreatitis on secretin magnetic resonance cholangiopancreatography
      * Abnormal endoscopic pancreatic function tests (peak HCO2 < 80mM)
    * Histopathology confirmed diagnosis of chronic pancreatitis
    * Compatible clinical history and documented hereditary pancreatitis gene mutation OR
    * History of recurrent acute pancreatitis (more than one episode of characteristic pain associated with imaging diagnostic of acute pancreatitis and/or elevated serum amylase or lipase > 3 times upper limit of normal
  * At least one of the following:

    * Daily narcotic dependence
    * Pain resulting in impaired quality of life, which may include: inability to attend school, recurrent hospitalizations, or inability to participate in usual, age-appropriate activities.
  * Complete evaluation with no reversible cause of pancreatitis present or untreated
  * Failure to respond to maximal medical and endoscopic therapy
* If clinical, radiologic, or biochemical evidence suggestive of cirrhosis or metabolic syndrome (defined in exclusion criteria), the participant has undergone hepatology evaluation and been exonerated of a cirrhosis diagnosis or otherwise deemed to be at low hepatic risk from IAT
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 2 years
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or active non-pancreatic malignancy are eligible for this trial
* Invasive abdominal surgical procedures such as pancreatectomy have the known potential to cause pregnancy loss. For this reason, persons of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to undergoing pancreatectomy and IAT. Should a participant become pregnant or suspect a pregnancy prior to planned pancreatectomy and IAT, the participant should inform their treating physician immediately

Exclusion Criteria:

* Prior allogenic or autologous islet cell transplantation
* Underlying liver disease, unless participant has undergone hepatology consultation to evaluate hepatic risk from IAT and been deemed low-risk, including:

  * Cirrhosis, defined by either

    * Pathologic diagnosis of cirrhosis OR
    * Diagnosis of cirrhosis by hepatology following evaluation prompted by clinical, radiographic, or biochemical evidence of cirrhosis
  * Hepatic steatosis as defined by pathologic examination of the liver or liver magnetic resonance imaging in the absence of pathologic evidence
* Use of any systemically absorbed steroid (e.g., prednisone but not budesonide) within the prior month
* Untreated malignancy of a non-pancreatic primary
* Cytology or biopsy of a pancreatic neoplasm diagnostic for malignancy prior to the time of IAT
* A pancreatic neoplasm deemed to be at high risk for harboring occult malignancy as assessed by the multi-disciplinary pancreas tumor board and multi-disciplinary chronic pancreatitis conference after comprehensive evaluation of relevant clinical, radiographic, pathologic, and serologic data. Features of high-risk neoplasms include the following, however the below items are not to be taken as absolute contraindications to TPIAT:

  * Obstructive jaundice in a patient with a pancreatic cystic neoplasm in the head of the pancreas
  * Enhancing mural nodule of any size
  * Main pancreatic duct >= 5mm
  * Acute pancreatitis with cystic lesion as the only potentially identifiable cause
  * Cyst >= 3cm, if lesion is a mucinous neoplasm
  * Thickened/enhancing cyst walls
  * Abrupt change in caliber of pancreatic duct with distal pancreatic atrophy on imaging
  * Celiac/portal lymphadenopathy
  * Serum CA19-9 above the institutional upper limit of normal
  * Pancreatic cyst growth rate >= 5mm every 2 years
  * Cytology suspicious for malignancy
  * Clinical suspicion for main duct involvement based on imaging
* Evidence of metabolic syndrome, as defined by any 3 of the below features, unless the participant has undergone hepatology consultation to evaluate hepatic risk from IAT and been deemed low-risk:

  * Waist circumference more than 40 inches in men and 35 inches in women
  * Elevated triglycerides 150 milligrams per deciliter of blood (mg/dL) or greater
  * Reduced high-density lipoprotein cholesterol (HDL) less than 40 mg/dL in men or less than 50 mg/dL in women
  * Elevated fasting glucose of 100 mg/dL or greater
  * Blood pressure values of systolic 130 mmHg or higher and/or diastolic 85 mmHg or higher
* Multifocal or large pancreatic neoplasms such that an insufficient volume of remnant pancreas would remain for the patient to benefit from IAT following resection of the neoplasms in the opinion of the multi-disciplinary chronic pancreatitis board
* History of allergic reaction to human albumin preparations
* Demonstrated medical non-compliance
* Patient unsafe to undergo the required pancreatectomy procedure in the opinion of the attending surgeon and/or anesthesiologist
* Patients deemed not suitable for the IAT follow-up protocol by any member of the multi-disciplinary IAT care team
* Any alcohol or tobacco use within 6 months of study enrollment
* Financial, logistic, or insurance constraints preventing adequate and timely pre-operative evaluation, case scheduling, or post-operative monitoring/follow-up
* Pregnant individuals are excluded from this study because invasive abdominal surgical procedures such as pancreatectomy have the known potential to cause pregnancy loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that are free of metastatic disease to the liver from a pancreatic primary | From date of surgery to time of identification of metastatic disease from a pancreatic primary, assessed up to 2 years post-surgery or date of death due to metastatic disease of a pancreatic origin
  The 95% confidence interval (CI) will be analyzed using the Clopper-Pearson exact interval method.

SECONDARY OUTCOMES:
Insulin free rate | From date of surgery to 2 years post-surgery or death by any cause
  Defined as proportion not requiring insulin for blood glucose control for at least 14 days prior to the assessment date at 2 years. The 95% CI will be analyzed using Clopper-Pearson exact interval method.
Opiates free rate | From date of surgery to 2 years post-surgery or death by any cause
  Defined as proportion not receiving opiates for at least 14 days prior to the assessment date at 2 years.The 95% CI will be analyzed using Clopper-Pearson exact interval method.
Time to overall survival (OS) | From date of surgery to 2 years post-surgery or death by any cause
  The time to OS distribution will be characterized using the Kaplan-Meier method. Kaplan-Meier curves of OS rate at 2 years will be estimated from the survival curve along with the 95% CI.

OTHER OUTCOMES:
Quality of life (QOL) | Up to 2 years
  QOL scores will be collected over time using the Short Form 12. Summary of QOL and its change over time will be presented graphically using box plot and spaghetti plots, in addition to a summary table of QOL over time.
Pain-related outcomes | Up to 2 years
  Subjective pain-related outcomes will be collected using Patient Reported Outcomes Measurement Information System Bank Pain Interference Survey, version 1.1 and will be analyzed similar to the QOL survey.
Incidence of adverse events (AEs) | Up to 2 years
  AEs of grade 3 or greater will be collected and tabulated by the Medical Dictionary for Regulatory Activities version 21.1. By-patient listings will also be provided for the following: patient deaths, serious adverse events, and AEs leading to withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Brett C Sheppard, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States